CLINICAL TRIAL: NCT02374541
Title: Screening and Linkage to Services for Autism
Acronym: SaLSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health and Hospital Authority (Other); Rocky Mountain Human Services (Other); El Grupo Vida (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 14-1728; R40MC27702 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2015-02-19; First posted 2015-03-02 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Autism Spectrum Disorders
Keywords: Patient Navigation; Health Disparities; Coordination of Services; Early Intervention (Education); Health Services Accessibility; Patient Advocacy
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Navigation (Experimental): Assistance from Autism Patient Navigator (APN) to obtain diagnostic evaluation / eligibility determination for possible autism spectrum disorder and, if indicated, early intervention services.
  Interventions: Behavioral: Patient Navigation
- Control (No Intervention): Standard referral for diagnostic evaluation / eligibility determination for possible autism spectrum disorder and, if indicated, early intervention services.

INTERVENTIONS:
Behavioral: Patient Navigation — The Autism Patient Navigator (APN) will interview families to determine system and individual barriers facing the family at each stage of the care process. The APN will help families to overcome any identified barriers through education, coaching, social support, interpretation or translation, linkage to resources (e.g., for obtaining insurance) or logistical support (e.g., scheduling appointments, providing reminders, arranging transportation), in order to ensure timely diagnostic evaluation / eligibility determination; educate the family about autism, tests and treatments; and offer psychosocial support.
  Other Names: Autism Patient Navigation
  Arms: Patient Navigation

SUMMARY:
The SaLSA (Screening and Linkage to Services for Autism) study will test whether patient navigation can help disadvantaged families obtain earlier diagnosis and treatment for their children who have had a positive screening test for autism spectrum disorder. Half of the families will be offered help from an autism patient navigator. The other half will receive standard care.

DETAILED DESCRIPTION:
Despite its relatively high rate of occurrence, autism spectrum disorder (ASD) is under-diagnosed and under-treated in young children, particularly in minority and disadvantaged populations. Although screening for ASD in the primary care setting is recommended as best practice, inadequate attention has been paid to addressing important obstacles to early recognition of ASD, including barriers to referral after positive screening, completion of diagnostic evaluations, and receipt of treatment. Patient navigation was originally developed to reduce health care disparities. The patient navigator guides patients with suspicious findings (e.g., a positive screening test) through and around barriers to care to ensure timely diagnosis and treatment. Patient navigation has improved receipt of preventive care among low-income, minority children but has not been tested for improving early identification and treatment of autism spectrum disorders. The goal of this study is to test the effectiveness and feasibility of patient navigation to facilitate autism screening follow-up, diagnostic evaluation, and linkage to early intervention in a very young, disadvantaged, minority population. To increase patient navigation's potential for widespread application and public health impact, this study uses the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework, a set of criteria for translating research into action, to guide planning and evaluation. The intervention's Reach, Effectiveness, Adoption, Implementation and Maintenance over time will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Receives medical care at Denver Community Health Services (DCHS) clinic
* Positive M-CHAT screening test (score 3 or higher) between ages 16 and 30 months at DCHS
* Resident of City and County of Denver

Exclusion Criteria:

* Existing diagnosis of autism spectrum disorder
* Sibling of enrolled subject

Ages: 16 Months to 32 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 305 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Completion of developmental evaluation / eligibility determination | 36 months of age
  Indicated developmental evaluation (aka eligibility determination) completed (Yes/No)

SECONDARY OUTCOMES:
Individualized Family Service Plan (IFSP) development | 36 months of age
  Documented development of indicated IFSP (Yes/No)
Age at Individualized Family Service Plan (IFSP) development | 36 months of age
  Age at indicated IFSP development (months)
Time to Individualized Family Service Plan (IFSP) development | 36 months of age
  Time from initial positive Modified Checklist for Autism in Toddlers, Revised (M-CHAT-R) screen to indicated IFSP development (days)
Initiation of indicated early intervention (EI) services | 36 months of age
  Initiation of at least one indicated EI service (Yes/No)
Age at initiation of indicated early intervention services | 36 months of age
  Age at initiation of any indicated EI service (months)
Time to initiation of indicated early intervention services | 36 months of age
  Time from initial positive Modified Checklist for Autism in Toddlers, Revised (M-CHAT-R) screen to initiation of any indicated EI service (days)
Referral for developmental evaluation / eligibility determination | 36 months of age
  Referral for developmental evaluation / eligibility determination made (yes/no)
Time to referral for and implementation of developmental evaluation / eligibility determination | 36 months of age
  Time from initial positive Modified Checklist for Autism in Toddlers, Revised with Follow-Up (M-CHAT-R/F screen to referral (days) and to completion of evaluation (days)
Age at referral for and implementation of developmental evaluation / eligibility determination | 36 months of age
  Age at referral (months) and age at completion of evaluation (months)

OTHER OUTCOMES:
Engagement in early intervention services for at least 3 months after initiation | 36 months of age
  At least one indicated early intervention service received 3 or more months after initiation of EI services (Yes/No)
Receipt of Modified Checklist for Autism in Toddlers, Revised (M-CHAT-R) Follow-up Interview | 36 months of age
  Receipt of indicated Modified Checklist for Autism in Toddlers, Revised with Follow-up (M-CHAT-R/F) (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn DiGuiseppi, MD, PhD, Principal Investigator — Colorado School of Public Health, University of Colorado Denver
Locations (3):
- United States (3):
  - Colorado School of Public Health, University of Colorado Denver, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No